CLINICAL TRIAL: NCT03092245
Title: Efficacy and Safety of OctaplasLG® Administration vs. Crystalloids (Standard) in Patients With Septic Shock - a Randomized, Controlled, Open-label Investigator-initiated Pilot Trial
Brief Title: Vasculopathic Injury and Plasma as Endothelial Rescue in Septic Shock (SHOCK) Trial
Acronym: VIPER-SHOCK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Octapharma (Industry); University of Iceland (Other)
Responsible Party: Principal Investigator, Jakob Stensballe, MD, PhD, Consultant Anaethetist, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: VIPER-SHOCK; 2017-000427-27 (EudraCT Number)
Record Dates: First submitted 2017-02-21; First posted 2017-03-27 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Ringer's acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OctaplasLG (Active Comparator): OctaplasLG® is an industrial donor plasma product pooled from 630 -1520 single donor units. It possesses unique features when compared to standard FFP, such as having a standardized concentration of natural pro- and anti-coagulation factors, a standardized volume as well as being pathogen-free.12 Most importantly, the manufacturing method of OctaplasLG® removes immune complexes and cells in several steps of microfiltration. The manufacturing process also inactivates viral, bacterial and prion pathogen by immune neutralization, solvent-detergent treatment and a prion specific ligand affinity chromatography step.
  Interventions: Drug: OctaplasLG
- Ringer-Acetate (Placebo Comparator): standard of care resuscitation fluid Ringer-acetate is a mixture of electrolytes in water to a slightly hypotonic solution.
  Interventions: Drug: Ringer-Acetate

INTERVENTIONS:
Drug: OctaplasLG — OctaplasLG is given as an infusion when resuscitation fluids are required.
  Other Names: Octaplas
  Arms: OctaplasLG
Drug: Ringer-Acetate — Ringer-acetate is given as an infusion when resuscitation fluids are required.
  Other Names: Ringer's Acetate
  Arms: Ringer-Acetate

SUMMARY:
Efficacy and safety of OctaplasLG® administration vs. crystalloids (standard) in patients with septic shock - a randomized, controlled, open-label investigator-initiated pilot trial

DETAILED DESCRIPTION:
This is a single center, randomized (1:1, active : standard of care), controlled, open-label, investigator-initiated pilot phase IIa trial in patients with septic shock investigating the efficacy and safety of administrating OctaplasLG® as compared to crystalloids, such as Ringer-Acetate (standard of care) in a total of 40 patients.

40 patients will be enrolled:

* Patients in the active treatment group (n = 20 patients) will receive OctaplasLG® as volume support according to trial algorithm.
* Patients in the standard of care group (n = 20 patients) will receive crystalloids, such as Ringer-Acetate, as volume support according to trial algorithm.

All patients will be treated according to the standard ICU care.

ELIGIBILITY:
Inclusion Criteria:

1. Adult intensive care patients (age ≥ 18 years) AND
2. Sepsis, defined as life-threatening organ dysfunction caused by a dysregulated host response to infection AND
3. Quick SOFA (qSOFA) with two or more of

   1. Respiratory rate ≥ 22/min
   2. Altered mentation (Glasgow Coma Scale score < 15)
   3. Systolic blood pressure ≤ 100mmHg AND
4. Septic shock, defined as a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP ≥65 mm Hg and having a serum lactate level >2 mmol/L despite adequate volume resuscitation AND
5. Requiring infusion of noradrenalin 0.10 mcg/kg/min or more to maintain blood pressure AND
6. Respiratory failure requiring intubation and mechanical ventilation

Exclusion Criteria:

1. Documented refusal of blood transfusion OR
2. Treatment with GPIIb/IIIa inhibitors < 24h from screening OR
3. Withdrawal from active therapy OR
4. Previously within 30 days included in an interventional trial OR
5. Known IgA deficiency with documented antibodies against IgA OR
6. Known hypersensitivity to OctaplasLG®: the active substance, any of the excipients (Sodium citrate dihydrate, Sodium dihydrogenphosphate dihydrate or Glycine) or residues from the manufacturing process (Tri (N-Butyl) Phosphate (TNBP) and Octoxynol (Triton X-100)) OR
7. Known severe deficiencies of protein S OR
8. Pregnancy (non-pregnancy confirmed by patient being postmenopausal or having a negative urine-hCG) OR
9. Severe cirrhotic hepatic failure with expected need for treatment with terlipressin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Microscan at 24 hours | 24 hours after baseline
  Change in microvascular perfusion from baseline to 24 hours after inclusion as evaluated by sidestream darkfield (SDF; MicroVision Medical, Amsterdam, The Netherlands) imaging technique.
Biomarkers at 24 hours | 24 hours after baseline
  Change in biomarkers indicative of endothelial activation and damage (sE-selectin, syndecan-1, thrombomodulin, VEGFR1, VEGF, nucleosomes) from baseline to 24 hours after inclusion.

SECONDARY OUTCOMES:
24 hour mortality | 24 hours after inclusion
  Difference in 24 hours mortality between patients receiving active treatment (OctaplasLG®) and standard of care (crystalloids such as Ringer-Acetate).
7 day mortality | 7 days after inclusion
  Difference in 7 day mortality between patients receiving active treatment (OctaplasLG®) and standard of care (crystalloids such as Ringer-Acetate).
30 day mortality | 30 days after inclusion
  Difference in 30 day mortality between patients receiving active treatment (OctaplasLG®) and standard of care (crystalloids such as Ringer-Acetate).
90 day mortality | 90 days after inclusion
  Difference in 90 day mortality between patients receiving active treatment (OctaplasLG®) and standard of care (crystalloids such as Ringer-Acetate).
Length of stay in the ICU | Days, assessed at 30-days and 90-days
  The number of days in the ICU after inclusion
Days on vasopressors | Days, assessed at 30-days and 90-days
  The number of days on vasopressors after inclusion
Days on ventilator | Days, assessed at 30-days and 90-days
  The number of days on vasopressors after inclusion
Transfusion requirements | For the first 7 days after inclusion
  Bleeding requiring > 2 RBC / day
Serious Adverse Reactions at 72 hours | For the first 72 hours after inclusion
  Severe adverse reactions, defined as symptomatic thromboembolism and TACO/TRALI
Serious Adverse Reactions at day 30 | At day 30 after inclusion
  Severe adverse reactions, defined as symptomatic thromboembolism and TACO/TRALI
Oxygenation | At 24 hours, 48 hours, 72 hours and at day 7 after baseline
  As evaluated by the PaO2/FiO2-ratio during the ICU stay
RIFLE criteria: Risk, Injury, and Failure, Loss and End-stage kidney disease | For the first 7 days in the ICU
  Acute Kidney Injury according to RIFLE criteria
Renal Replacement Therapy | For the first 7 days after inclusion
  recording whether the patient is receiving dialysis or not

OTHER OUTCOMES:
Sepsis-related organ failure assessment (SOFA) | At 24 hours, 48 hours, 72 hours and at day 7 after baseline
  Worst score in a 24 hour period
Thrombelastograph (TEG) maximum amplitude at 24 hours | At 24 hours after baseline
  Measuring the maximum amplitude (MA) in mm with TEG
Thrombelastograph (TEG) maximum amplitude at 48 hours | At 48 hours after baseline
  Measuring the maximum amplitude (MA) in mm with TEG
Thrombelastograph (TEG) maximum amplitude at 72 hours | At 72 hours after baseline
  Measuring the maximum amplitude (MA) in mm with TEG
Thrombelastograph (TEG) Functional Fibrinogen maximum amplitude at 24 hours | At 24 hours after baseline
  Measuring the maximum amplitude (MA) in mm with TEG Functional Fibrinogen (FF)
Thrombelastograph (TEG) Functional Fibrinogen maximum amplitude at 48 hours | At 48 hours after baseline
  Measuring the maximum amplitude (MA) in mm with TEG Functional Fibrinogen (FF)
Thrombelastograph (TEG) Functional Fibrinogen maximum amplitude at 72 hours | At 72 hours after baseline
  Measuring the maximum amplitude (MA) in mm with TEG Functional Fibrinogen (FF)
Disseminated Intravascular Coagulation (DIC) score | At 24 hours, 48 hours, 72 hours and at day 7 after baseline
  Total score in a 24 hour period based upon platelets, INR, Fibrinogen and D-dimer lab results.

CONTACTS AND LOCATIONS:
Overall Officials: Niels E Clausen, Principal Investigator — Bispebjerg and Frederiksberg Hospitals, Capitol Region of Copenhagen
Locations (1):
- ICU Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No